CLINICAL TRIAL: NCT04452149
Title: Algorithm Using LINQ Sensors for Evaluation And Treatment of Heart Failure
Acronym: ALLEVIATE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALLEVIATE-HF
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: Heart Failure; Insertable Cardiac Monitor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Following Reveal LINQ™ device insertion, subjects will be randomly allocated in a blinded fashion in a 1:1 ratio to either the observation arm or the intervention arm. Subjects in the observation arm will start with an observational period of 13 months and then transition to the intervention arm for the remainder of their participation in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study site personnel and subjects will remain blinded to the subject's randomization assignment until the 13-month timepoint at which point the subjects will be in the intervention arm for the remainder of their participation regardless of original allocation, or until the time of investigator and/or subject contact in relation to a "high" risk status in an intervention arm subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Observation Arm (Placebo Comparator): Subjects will receive a Reveal LINQ™ Insertable Cardiac Monitor with an investigational ALLEVIATE-HF RAMware download, and will be managed per standard of care for heart failure management without visibility to the heart failure sensor data. Subjects will transition to the intervention arm after 13 months.
  Interventions: Device: Reveal LINQ™ Insertable Cardiac Monitor with investigational ALLEVIATE-HF RAMware download
- Intervention Arm (Experimental): Subjects will receive a Reveal LINQ™ Insertable Cardiac Monitor with an investigational ALLEVIATE-HF RAMware download, and will be managed using an integrated device diagnostic-based risk stratification algorithm combined with a clinical medication plan.
  Interventions: Device: Reveal LINQ™ Insertable Cardiac Monitor with investigational ALLEVIATE-HF RAMware download; Other: Medication intervention

INTERVENTIONS:
Device: Reveal LINQ™ Insertable Cardiac Monitor with investigational ALLEVIATE-HF RAMware download — Reveal LINQ™ Insertable Cardiac Monitor with investigational ALLEVIATE-HF RAMware download.
Other: Medication intervention — Risk status guided medication intervention.
  Arms: Intervention Arm

SUMMARY:
The ALLEVIATE-HF study is a prospective, randomized, controlled, blinded, multi-site, interventional, investigational device exemption (IDE) pivotal study. The purpose of the study is to demonstrate the safety and efficacy of a patient management pathway that utilizes an integrated device diagnostic-based risk stratification algorithm to guide patient care in subjects with NYHA class II and III heart failure, and to demonstrate the safety of the Reveal LINQ™ system and procedure in the study population.

DETAILED DESCRIPTION:
The study will utilize the market released Reveal LINQ™ Insertable Cardiac Monitor with an investigational ALLEVIATE-HF RAMware download. The study will enroll up to 900 subjects at up to 75 sites in the US. Subjects will be followed until the last enrolled subject is followed for 7 months or until the end of the study, whichever occurs first, or until time of study exit or death as applicable, but no longer than 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has NYHA Class II or III heart failure per most recent assessment, irrespective of left ventricular ejection fraction (LVEF)
* Patient has documented recent history of symptomatic heart failure, defined as meeting any one of the following three criteria: 1. Hospital admission with primary diagnosis of HF within the last 12 months, OR 2. Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration within the last 6 months, OR 3. Patient had the following BNP/NT-proBNP within the last 3 months: If LVEF ≥ 50%, then BNP> 150 pg/ml or NT-proBNP > 450 pg/ml OR If LVEF is <50%, then BNP> 300 pg/ml or NT-proBNP > 900 pg/ml
* Patient is willing and able to comply with the protocol, including LINQ ICM insertion, CareLink transmissions (including adequate connectivity), study visits and remote care directions.
* Patient is 18 years of age or older.
* Patient has a life expectancy of 12 months or more.

Exclusion Criteria:

* Patient is currently implanted with a cardiovascular implantable electronic device (CIED) (e.g. ICM, pacemaker, ICD, CRT-D or CRT-P device) or hemodynamic monitor.
* Patient is receiving temporary or permanent mechanical circulatory support.
* Patient had MI or PCI/CABG within past 90 days.
* Patient has had a heart transplant, or is currently on heart transplant list.
* Patient has severe valve stenosis on echocardiogram.
* Patient has primary pulmonary hypertension (pre-capillary, WHO group 1,3,4,5).
* Patient is on chronic intravenous inotropic drug therapy (e.g. dobutamine, milrinone).
* Patient has severe renal impairment (eGFR <30 mL/min).
* Patient has systolic blood pressure of < 90 mmHg at the time of enrollment.
* Patient is on chronic renal dialysis.
* Patient is unable to undergo one round of PRN medication intervention (i.e. 4 days of increased diuretics dose).
* Patient has liver disease, defined as AST/ALT >5x normal, or bilirubin >2x normal.
* Patient has serum albumin < 3 g/dL.
* Patient has hypertrophic obstructive cardiomyopathy, constrictive pericarditis or amyloidosis.
* Patient has complex adult congenital heart disease.
* Patient has active cancer involving chemotherapy and/or radiation therapy.
* Patient weighs more than 500 pounds.
* Patient is pregnant or breastfeeding (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment).
* Patient is enrolled in another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Safety of patient management pathway - Proportion of medication interventions with associated medication intervention related serious adverse events | Up to 3 years
  The proportion of medication interventions with one or more associated medication intervention related SAEs will be evaluated.
Efficacy of patient management pathway - Hierarchical composite of Cardiovascular death, HF events, change in Kansas City Cardiomyopathy Questionnaire and change in six-minute walk test distance | Follow-up duration at endpoint analysis ranges from a minimum of 7 to a maximum of 13 months
  Treatment and Control groups will be compared using the Finkelstein-Schoenfeld method, including subjects with at least one "high" heart failure risk status.

SECONDARY OUTCOMES:
Safety of Reveal LINQ™ system and procedure - Percentage of subjects experiencing system or procedure related serious adverse events | Up to 6 months post Reveal LINQ™ device insertion attempt
  Freedom from Reveal LINQ™ system and procedure related serious adverse events at 6 months will be evaluated.
Efficacy of patient management pathway - Hierarchical composite of Cardiovascular death, HF events, change in Kansas City Cardiomyopathy Questionnaire, change in six-minute walk test distance, and change in device-measured activity and night heart rate | Follow-up duration at endpoint analysis ranges from a minimum of 7 to a maximum of 13 months
  Treatment and Control groups will be compared using the Finkelstein-Schoenfeld method, including subjects with at least one "high" heart failure risk status.

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, Principal Investigator — Baylor Scott and White Health
Locations (53):
- United States (53):
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Saint Joseph Heritage Healthcare, Mission Viejo, California
  - Cardiology Associates Medical Group, Oxnard, California
  - Saint Joseph's Medical Center, Stockton, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - FWD Clinical Research LLC, Boca Raton, Florida
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Florida Heart Center, Ft. Pierce, Florida
  - Baptist Health, Jacksonville, Florida
  - First Coast Cardiovascular Institute PA, Jacksonville, Florida
  - Citrus Cardiology Consultants PA, Leesburg, Florida
  - Baptist Hospital, Pensacola, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - NorthShore University Health System, Evanston, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Parkview Health, Fort Wayne, Indiana
  - Ascension Medical Group - Saint Vincent, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Healthcare System, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - North Memorial Health Heart & Vascular Center, Robbinsdale, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - CHI Health Creighton University Medical Center - Bergan Mercy, Omaha, Nebraska
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New Mexico Heart Institute PA, Albuquerque, New Mexico
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Saint Francis Hospital, Roslyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Cone Health, Greensboro, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - Mount Carmel East, Columbus, Ohio
  - OhioHealth Research and Innovation Institute (OHRI), Columbus, Ohio
  - Doylestown Health Cardiology a division of Doylestown Health Physicians, Doylestown, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands, Columbia, South Carolina
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - University of Tennessee Methodist Physicians, Memphis, Tennessee
  - Medical City Fort Worth, Fort Worth, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center Cherry Hill, Seattle, Washington
  - Saint Joseph Medical Center (Tacoma WA), Tacoma, Washington
  - Charleston Area Medical Center (CAMC) Memorial Hospital, Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahwash R, Zile MR, Chalasani P, Bertolet B, Gravelin L, Khan MS, Wehking J, Van Dorn B, Sarkar S, Laager V, Gerritse B, Laechelt A, Butler J; ALLEVIATE-HF Phase I Investigators. Personalized Intervention Strategy Based on a Risk Score Generated From Subcutaneous Insertable Cardiac Monitor: Results From Phase 1 of ALLEVIATE-HF. J Am Heart Assoc. 2024 Oct 15;13(20):e035501. doi: 10.1161/JAHA.124.035501. Epub 2024 Oct 11. PMID 39392161
- [Derived] Zile MR, Kahwash R, Sarkar S, Koehler J, Zielinski T, Mehra MR, Fonarow GC, Gulati S, Butler J. A Novel Heart Failure Diagnostic Risk Score Using a Minimally Invasive Subcutaneous Insertable Cardiac Monitor. JACC Heart Fail. 2024 Jan;12(1):182-196. doi: 10.1016/j.jchf.2023.09.014. Epub 2023 Nov 8. PMID 37943225